CLINICAL TRIAL: NCT06291064
Title: TreAtment Response and Omic-Markers in Triple-Negative Breast CAncer Patients Receiving Standard of Care Chemotherapy (TARMAC)
Brief Title: Trial Studying Chemotherapy in Nigerian Women With Triple Negative Breast Cancer
Acronym: TARMAC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0678
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Docetaxel; Carboplatin; Mastectomy, Segmental; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Participants will receive epirubicin and cyclophosphamide every three weeks for a total of 12 weeks followed by 3-weekly docetaxel for 12 weeks and carboplatin every three weeks for a total of 12 weeks. All premenopausal participants will receive luteinizing hormone-releasing hormone (LHRH) agonist goserelin (Zoladex) for contraception and fertility preservation.
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Docetaxel; Drug: Carboplatin; Procedure: Breast Surgery; Drug: Capecitabine

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide is given by intravenous (IV) infusion once every 3 weeks for 4 doses total (12 weeks). It will be given together with Epirubicin.
Drug: Epirubicin — Epirubicin is given by intravenous (IV) infusion once every 3 weeks for 4 doses total (12 weeks). It will be given together with Cyclophosphamide.
Drug: Docetaxel — Docetaxel is given by intravenous (IV) infusion once every 3 weeks for 4 doses total (12 weeks). It will be given together with Carboplatin. Dosing will start after treatment with Epirubicin and Cyclophosphamide (EC) is completed.
Drug: Carboplatin — Carboplatin is given by intravenous (IV) infusion once every 3 weeks for 4 doses total (12 weeks). It will be given together with Docetaxel. Dosing will start after treatment with EC is completed.
Procedure: Breast Surgery — Participants will undergo breast surgery after completing dosing with Carboplatin and Docetaxel to remove any remaining cancer in the breast.
Drug: Capecitabine — Capecitabine is a pill that will be taken by mouth daily for 6 months after surgery is completed.

SUMMARY:
The primary purpose of this study is to determine what proportion of participants will achieve complete pathological response with epirubicin+ cyclophosphamide followed by docetaxel +carboplatin. This will also examine the potential of using signals in the blood (biomarkers) to identify resistance to chemotherapy in Nigerian women with triple negative breast cancer (TNBC).

All enrollment to this trial will occur at sites in Nigeria. University of Chicago is serving as coordinating center and will be involved in data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages of 18 to 70 years old
2. Women who are able and willing to read understand and sign an informed consent document
3. Biopsy-accessible breast tumor of significant size for core needle biopsy/ultrasound measurable (≥ 2cm)
4. Patients with histologically confirmed carcinoma of the female breast with triple-negative status by immunohistochemistry (IHC). Patients who are low estrogen reception (ER) expression (< 20%), progesterone receptor (PR) negative and human epidermal growth factor 2 (HER2) negative are eligible.
5. Clinical stages IIA -IIIC (AJCC 2009)
6. Chemotherapy-naïve patients (for this cancer)
7. Performance status: Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Non-pregnant and not nursing.

   * Granulocyte greater than or equal to 1,500/microliter
   * Platelet count greater than or equal to 100,000/microliter
   * Absolute neutrophil count (ANC) greater than or equal to l500/microliter
   * Hemoglobin greater than or equal to 10g/deciliter
   * Bilirubin less than or equal 1.5 x upper limit of normal
   * aspartate aminotransferase (ALT or SGOT) and alanine transaminase (AST or SGPT) less than 2.5 x upper limit of normal

7. Creatinine within institutional normal limits or glomerular filtration rate greater than or equal to 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation 10. Baseline left ventricular ejection fraction of greater than or equal to 55%

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with distant metastasis (brain and/or visceral metastasis)
3. Serious, uncontrolled, concurrent infection(s).
4. Treatment for other carcinomas within the last 5 years, except non-melanoma skin cancer and treated cervical carcinoma in-situ (CCIS)
5. Participation in any investigational drug study within 4 weeks preceding the start of study treatment
6. Other serious uncontrolled medical conditions that the treating investigator feels might compromise study participation including but not limited to chronic or active infection, HIV-positive patient, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study will enroll women with breast cancer.
Enrollment: 85 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that Achieve Pathologic Complete Response (pCR) Rate (Breast) | 4 - 6 months from start of chemotherapy
  How well does the study chemotherapy regimen of epirubicin and cyclophosphamide (EC) followed by docetaxel and carboplatin work to remove tumor cells in the breast. This will be determined by percentage of participants that do not have noticeable cancer cells in the breast after completing the chemotherapy regimen.
Percentage of Participants that Achieve Pathologic Complete Response (pCR) Rate (Lymph Nodes) | 4 - 6 months from start of chemotherapy
  How well does the study chemotherapy regimen of epirubicin and cyclophosphamide (EC) followed by docetaxel and carboplatin work to remove tumor cells in the lymph nodes. This will be determined by percentage of participants that do not have noticeable cancer cells in the lymph nodes after completing the chemotherapy regimen.
Percentage of Participants that Achieve Pathologic Complete Response (pCR) Rate (By Stage) | 4 - 6 months from start of chemotherapy
  How well does the study chemotherapy regimen of epirubicin and cyclophosphamide (EC) followed by docetaxel and carboplatin work to remove tumor cells based on stage of breast cancer. This will be determined by percentage of participants that do not have noticeable cancer cells in the lymph nodes after completing the chemotherapy regimen.

SECONDARY OUTCOMES:
Side Effects of the Study Pre-surgery Chemotherapy Regimen | After 8 cycles of treatment (24 weeks)
  Percentage of participants experiencing Grades 3 and 4 blood, gastrointestinal, neurological and cardiovascular toxicities.
Clinical Response | 4 - 6 months from start of chemotherapy
  Percentage of participants achieving clinical response (CR and PR) during neoadjuvant period by breast ultrasound
Progressive Disease | After 8 cycles of treatment (24 weeks)
  Percentage of participants with progressive disease during pre-surgery treatment period
Invasive Disease Free Survival (iDFS) | 10 years from start of treatment
  Time to cancer returning or death
Duration of Response | 10 years from start of treatment
  Time to cancer worsening or death
Heart Related Side Effects of the Pre-Surgery Chemotherapy Regimen | 10 years from start of treatment
  Percentage of participants with Heart failure (NYHA Class III or IV or as confirmed by a cardiologist) and a decrease in left ventricular ejection fraction (LVEF) of at least 10 ejection fraction (EF) points from baseline and to below 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo Olopade, MD, Study Chair — University of Chicago
Locations (4):
- Nigeria (4):
  - Lagos State University Teaching Hospital, Ikeja, Lagos
  - Lagos University Teaching Hospital, Yaba, Lagos
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State
  - University of Ibadan Hospital, Ibadan, Oyo State